CLINICAL TRIAL: NCT02797418
Title: "Cognitus & Moi": a New Cognitive Remediation Tool for Children With Intellectual Deficiency With Behavioral Disorders
Brief Title: "Cognitus & Moi": a New Cognitive Remediation Tool
Acronym: COGNITUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-A00858-41
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Mental Retardation
Keywords: Attentional disorders, intellectual deficiency
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitus and Me (Experimental): Cognitus & Me is a cognitiv remediation program focused on the functions of attention and visuospatial that is to say that can move in space, to perceive objects of our environment and organize them, to mentally imagine a physically absent operation object very involved in social behavior, in order to limit the presence of behavioral disorders among children with intellectual disabilities.
  Interventions: Behavioral: Cognitive remediation program
- control group (Active Comparator): the control management that involves fine motor skills and research computer information,management control is usually done
  Interventions: Behavioral: Cognitive remediation program

INTERVENTIONS:
Behavioral: Cognitive remediation program — Comparison between a cognitive remediation program (Cognitus and Me") (groupe 1) and a training group of fine motor skills (group 2)

SUMMARY:
Holders children with intellectual disabilities have great difficulty in adapting to social situations and relationships.Cognitive impairment associated with intellectual disability are important factors to understand their difficulties in processing social information. In the field of recognition of facial emotions in particular, basic cognitive processes such as visuospatial and attentional functions, are heavily involved.Cognitive remediation is a management tool widely used by practitioners to help patients who experience cognitive difficulties. Currently, no program can meet specific and validated the problems are children with intellectual disabilities manner in their daily functioning.

DETAILED DESCRIPTION:
Cognitus & ME is a remediation program focused on attentional functions and visuospatial, to limit the presence of behavioral disorders among children with intellectual disabilities.The main objective is to validate the effectiveness of Cognitus & ME program on behavioral disorders in children with intellectual disabilities (with or without autism spectrum disorder associated).

ELIGIBILITY:
Inclusion Criteria:

* Children with intellectual deficiency (5-13 years) (40 < total IQ < 75) with or without autism spectrum disorders
* Native French speaker
* Clinically stable
* Parental consent

Exclusion Criteria:

* visual or auditory disorder
* history of neurological illness or trauma
* Absence of language

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist scale | 6 months
  Change in sub-score " hyperactivity / non compliance " (scale " Aberrant Behavior Checklist ") (completed by parents or the educational team). This measure is repeated at the end of the intervention to highlight the impact of the " Cognitus and Me " program, and 6 months later to investigate the possible long-lasting effects of the benefits.

SECONDARY OUTCOMES:
MDI-C scale ( Multiscore Depression Inventory for Children scale) | 6 months
  The Aberrant Behavior Checklist-Community (ABC-C; Aman & Singh, 1994) is a rating scale that measures the severity of a range of problem behaviors commonly observed in individuals with intellectual and developmental disabilities
KIDSCREEN-27 scale | 6 months
  The KIDSCREEN-27 with five dimensions resulted. All five dimensions are Rasch scales: Physical Well-Being (5 items), Psychological Well-Being (7 items), Autonomy & Parents (7 items), Peers & Social Support (4 items), and School Environment (4 items).
Vineland 2 scale (Vineland Adaptive Behavior Scale) | 6 months
  A measure of adaptive behavior from birth to adulthood
ABC scale (Irritability and social withdrawal) | 6 months
  This measure is repeated at the end of the intervention to highlight the impact of the " Cognitus and Me " program, and 6 months later to investigate the possible long-lasting effects of the benefits

CONTACTS AND LOCATIONS:
Overall Officials: DEMILY DR CAROLINE, MD PH, Principal Investigator — Le Vinatier Hospital
Locations (1):
- Demily Caroline, Bron, LYON, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Favre E, Peyroux E, Babinet MN, Poisson A, Demily C. Computer-based cognitive remediation program for the treatment of behavioral problems in children with intellectual disability: the <<COGNITUS & MOI>> study protocol for a randomized controlled trial. BMC Psychiatry. 2018 Jul 20;18(1):235. doi: 10.1186/s12888-018-1810-z. PMID 30029627